CLINICAL TRIAL: NCT04917497
Title: Levosimendan Infusion in Critically Ill Patients With Cardiogenic Shock
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: Levosimendan
Record Dates: First submitted 2021-05-31; First posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-06

CONDITIONS: Cardiogenic Shock; Cardiorenal Syndrome; Acute Kidney Failure
Keywords: Levosimendan; Inotropic Agent
MeSH Terms: conditions — Shock, Cardiogenic; Cardio-Renal Syndrome; Acute Kidney Injury | interventions — Simendan

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Levosimendan Treated Group: All patients consecutively admitted to the medical ICU of the University Hospital Zurich aged over 18 years, with an underlying cardiogenic shock, receiving Levosimendan.
  Interventions: Drug: Levosimendan

INTERVENTIONS:
Drug: Levosimendan — Levosimendan was administered according to a standardized treatment protocol. A total dose of 12.5mg or 25mg (corresponding to one or two ampoules) was given at an infusion rate of 0.05 μg/kg/min to 0.2μg/kg/min with or without a loading dose (6 μg/kg or 3 μg/kg over 10 minutes). The decision about total dose, infusion rate and loading dose was at the discretion of the treating physician.

SUMMARY:
To determine whether Levosimendan infusion in patients with cardiogenic shock and cardiorenal syndrome refractory to standard inotropic therapy, improves hemodynamics and renal function, whilst being safe.

DETAILED DESCRIPTION:
Cardiogenic Shock or the state of systemic hypoxia albeit initially preserved intra-vascular volume and intact vascular function, is solely the result of insufficient cardiac output [1-2]. The ensuing centralization and redistribution of blood-volume, is induced by a stimulation of the renin-angiotensin system, as well as vasopressin and endogenous catecholamine liberation [2-3]. Precipitating Cardiogenic Shock has a direct effect on the kidney, also called the cardiorenal syndrome [4].

The overall consensus for the therapy of cardiogenic shock is the use of inotropes to increase cardiac output and reverse organ hypoxia [2], nevertheless their increase of myocardial and glomerular oxygen consumption make them a double edged sword to use in cardiogenic shock and more prominently in cardiogenic shock coupled with pronounced cardiorenal syndrome.

Levosimendan is an inotropic agent that was developed for the treatment of severely decompensated heart failure. It exerts its inotropic effects primarily through sensitizing Troponin C to calcium and thereby increasing contraction of cardiac myofilaments during systole [5]. Unlike other inotropic agents, Levosimendan acts independently of the beta adrenergic receptor [5]. Additionally, the effect of Levosimendan could be beneficial for the kidneys function by decreasing pre-glomerular arteriolar vasotonus whilst keeping post-glomerular arteriolar vasotonus constant [6].

In light of the scarce but promising literature the question arises if Levosimendan can safely ameliorate cardiac and renal function concomitantly in patients presenting the combination of cardiogenic shock and cardiorenal syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Levosimendan
* Cardiogenic Shock
* Continuous monitoring of cardiac output at the start of and during treatment with Levosimendan

Exclusion Criteria:

* Extracorporal hemodynamic support or an implanted ventricular assist device
* Previous therapy with Levosimendan during the index hospitalization
* Refusal of participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients consecutively admitted to the medical ICU of the University Hospital Zurich aged over 18 years, with an underlying cardiogenic shock, receiving Levosimendan
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2011-06-30 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Cardiac Index | Mixed Model Assessment at 0, 1, 2, 4, 6, 12, 24, 48, 72, 96 and 120 hours post Levosimendan Infusion
  Temporal development of Cardiac Index post Levosimendan Infusion up until 120 hours
Change in Cardiac Preload Pressures | Mixed Model Assessment at 0, 1, 2, 4, 6, 12, 24, 48, 72, 96 and 120 hours post Levosimendan Infusion
  Temporal development of Wedge Pressure/ Central Venous Pressure post Levosimendan Infusion up until 120 hours
Change in Mean Arterial Pressure | Mixed Model Assessment at 0, 1, 2, 4, 6, 12, 24, 48, 72, 96 and 120 hours post Levosimendan Infusion
  Temporal development of Mean Arterial Pressure post Levosimendan Infusion up until 120 hours
Change in Vasoactive/ Inotropic Dosage | Mixed Model Assessment at 0, 1, 2, 4, 6, 12, 24, 48, 72, 96 and 120 hours post Levosimendan Infusion
  Temporal development of Norepinephrine/ Dobuatmine Dosage post Levosimendan Infusion up until 120 hours
Change in Renal Function | Mixed Model Assessment at 0, 1, 2, 4, 6, 12, 24, 48, 72, 96 and 120 hours post Levosimendan Infusion
  Temporal development of eGFR (Creatinin estimated) post Levosimendan Infusion up until 120 hours
Change in Fluid Balance | Mixed Model Assessment at 0, 1, 2, 4, 6, 12, 24, 48, 72, 96 and 120 hours post Levosimendan Infusion
  Temporal development of Fluid Balance post Levosimendan Infusion up until 120 hours

CONTACTS AND LOCATIONS:
Overall Officials: Marco Maggiorini, Principal Investigator — Medizinische Intensivstation D-HOER 27, UniversitatsSpital Zürich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Califf RM, Bengtson JR. Cardiogenic shock. N Engl J Med. 1994 Jun 16;330(24):1724-30. doi: 10.1056/NEJM199406163302406. No abstract available. PMID 8190135
- [Background] van Diepen S, Katz JN, Albert NM, Henry TD, Jacobs AK, Kapur NK, Kilic A, Menon V, Ohman EM, Sweitzer NK, Thiele H, Washam JB, Cohen MG; American Heart Association Council on Clinical Cardiology; Council on Cardiovascular and Stroke Nursing; Council on Quality of Care and Outcomes Research; and Mission: Lifeline. Contemporary Management of Cardiogenic Shock: A Scientific Statement From the American Heart Association. Circulation. 2017 Oct 17;136(16):e232-e268. doi: 10.1161/CIR.0000000000000525. Epub 2017 Sep 18. PMID 28923988
- [Background] Hochman JS. Cardiogenic shock complicating acute myocardial infarction: expanding the paradigm. Circulation. 2003 Jun 24;107(24):2998-3002. doi: 10.1161/01.CIR.0000075927.67673.F2. No abstract available. PMID 12821585
- [Background] Ronco C, House AA, Haapio M. Cardiorenal syndrome: refining the definition of a complex symbiosis gone wrong. Intensive Care Med. 2008 May;34(5):957-62. doi: 10.1007/s00134-008-1017-8. Epub 2008 Feb 5. PMID 18251008
- [Background] Papp Z, Edes I, Fruhwald S, De Hert SG, Salmenpera M, Leppikangas H, Mebazaa A, Landoni G, Grossini E, Caimmi P, Morelli A, Guarracino F, Schwinger RH, Meyer S, Algotsson L, Wikstrom BG, Jorgensen K, Filippatos G, Parissis JT, Gonzalez MJ, Parkhomenko A, Yilmaz MB, Kivikko M, Pollesello P, Follath F. Levosimendan: molecular mechanisms and clinical implications: consensus of experts on the mechanisms of action of levosimendan. Int J Cardiol. 2012 Aug 23;159(2):82-7. doi: 10.1016/j.ijcard.2011.07.022. Epub 2011 Jul 23. PMID 21784540
- [Background] Bragadottir G, Redfors B, Ricksten SE. Effects of levosimendan on glomerular filtration rate, renal blood flow, and renal oxygenation after cardiac surgery with cardiopulmonary bypass: a randomized placebo-controlled study. Crit Care Med. 2013 Oct;41(10):2328-35. doi: 10.1097/CCM.0b013e31828e946a. PMID 23921271